CLINICAL TRIAL: NCT01211496
Title: High Velocity Resistance Training in Older Men and Women
Brief Title: The Effect of Velocity Training in Functionally Limited Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 1042318; R03AG025141-01 (NIH)
Record Dates: First submitted 2008-12-02; First posted 2010-09-29 (Estimated); Last update posted 2016-10-04 (Estimated); Status verified 2016-10

CONDITIONS: Aging
Keywords: functional testing; resistance training; velocity training; elderly; geriatric; knee; leg; leg strength
MeSH Terms: interventions — Resistance Training

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- High-speed power training (Active Comparator): Volunteers randomized into High-speed power training (HSPT) will be exercised 3 times per week for 12 weeks. Each training session will consist of 3 sets of 12 to 14 repetitions at 40% of maximal strength for leg press (LP) and seated knee extension (KE) exercises.
  Interventions: Behavioral: High-speed power training
- Slow-speed strength training (Active Comparator): Volunteers randomized into Slow-speed strength training (SSST) will be exercised 3 times per week for 12 weeks. Each training session will consist of 3 sets of 8 to 10 repetitions at 80% of maximal strength for LP and KE exercises.
  Interventions: Behavioral: Slow-speed strength training
- placebo exercise (control group) (No Intervention): Volunteers randomized into the control group (CON) will undergo a placebo exercise intervention consisting of lower extremity range of motion and flexibility exercises performed 2 times per week with the assistance of the research staff.

INTERVENTIONS:
Behavioral: High-speed power training — High speed resistance training, 3 sessions per week for 12 weeks
  Other Names: power training; weight training
  Arms: High-speed power training
Behavioral: Slow-speed strength training — Slow speed resistance training, 3 sessions per week for 12 weeks
  Other Names: weight training
  Arms: Slow-speed strength training

SUMMARY:
We are exploring a unique weight-training program for men and women 65 years or older that emphasizes high speed training. We believe that the speed at which muscles move may be more important to the performance of functional tasks than how strong the muscles are. We are comparing velocity training with traditional strength training to determine which method has the greatest effects on muscle strength, speed of movement, functional performance and physical disability. We believe that higher speed training will improve these measures to a greater extent than simply training for increased muscle strength.

Aging also results in loss of bone mass, which increases the risk for falls and fractures. Strength training also has been shown to maintain bone mass in the elderly, but no studies have examined high velocity resistance training and maintenance of bone mass. We believe it is important to examine this aspect of velocity training before recommendations can be made.

DETAILED DESCRIPTION:
The study compared 12 weeks of explosive high-speed power training with traditional slow-speed strength training. Outcome measures included muscle performance: leg press (LP) and knee extension (KE) one-repetition maximum (1RM) and LP peak power (PP), velocity at peak power (PPV) and force at peak power (PPF) from 40%-90% of the 1RM. Measures of function consisted of habitual and maximal gait velocity, the short physical performance battery (SPPB), forward tandem walk, and lower limb movement time (braking speed) on an automobile driving simulator.

Participants reported to the laboratory for 2 weeks of baseline measurements. On visit 1, subjects were explained the study and completed an informed consent document. On visit 2 and 3, muscle performance and functional measures were obtained. The following week, all muscle performance and functional measures were repeated to establish reliability. At the end of baseline testing, participants were randomized to treatment. Following the 12-week RT intervention, post-training muscle performance and functional measures were obtained.

Resistance Training Protocol. Volunteers randomized into high-speed power training (HSPT) and slow-speed strength training (SSST) exercised 3 times per week for 12 weeks using computer-interfaced Keiser a420 pneumatic leg press and knee extension RT equipment (Fresno, CA). For HSPT, each training session consisted of 3 sets of 12-14 repetitions at 40%1RM. Participants performed an explosive movement at high speed during the concentric phase of each repetition, paused for one-second, and performed the eccentric portion of the contraction over 2 seconds. Volunteers randomized into SSST also exercised 3 times per week for 12 weeks with each training session consisting of 3 sets of 8-10 repetitions at 80%1RM. The participants performed each movement at a slow velocity (2 s for concentric phase of the repetition), paused for one second, and performed the eccentric portion of the contraction over 2 seconds. CON met three times a week for warm-up and stretching exercises, but performed no RT. HSPT and SSST participated in the same warm-up and stretching exercises as CON.

Measures Maximal strength and power. Leg press and seated knee extension 1RM were obtained using Keiser pneumatic RT equipment fitted with a420 electronics. The seat of both the recumbent LP and KE apparatus was positioned to place the hip and knee joints between 90 and 100 degrees of flexion. The 1RM was obtained by progressively increasing resistance until the subject was no longer able to push out one repetition successfully. The Borg Scale was used to assist in evaluating when 1RM (combined with perceived maximal effort) was reached. Peak muscle power was obtained at 40%, 50%, 60%, 70%, 80% and 90% of the 1RM approximately 30 minutes after 1RM testing (8,9). Participants were instructed to exert "as fast as possible" at each relative percentage of the 1RM. Three attempts were made at each resistance and the greatest PP output obtained at each resistance was used in the analysis. The corresponding PPV and PPF were obtained for each external resistance from 40%-90% 1RM. The 1RM was measured bi-weekly in HSPT and SSST only and relative training intensity was adjusted accordingly to ensure adequate overload during training. Post-training muscle performance measures were obtained using loads relative to the initial baseline 1RM as well as the post-training 1RM.

ELIGIBILITY:
Inclusion Criteria:

* 65 years of age
* relatively inactive
* male or female
* good overall health
* living independently (not in a nursing home or care facility)

Exclusion Criteria:

* physically active/athletic
* heart attack or unstable angina within 6 months of consent
* hip fracture, knee or hip replacement within 6 months of consent
* diagnosed neurological disease
* pulmonary disease requiring use of oxygen
* osteoarthritis of the knee
* severe visual or hearing impairment

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 52 (Actual)
Dates: Start 2004-06; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Strength and Power | 6 months
  The strength and power of the lower limb muscles will be measures using Keiser pneumatic leg press and knee extension exercise machines. The Keiser machines allow for the specific measurement of the contributions of force and velocity to the development of power, which will reveal whether the high-speed training protocol impacts speed-related measures of muscle performance.

SECONDARY OUTCOMES:
Mobility and Function | 6 months
  Walking speed tests (habitual gait speed and maximal gait speed), balance (tandem walk), stair climbing performance, chair rise time, and the timed up and go test will be used as overall measures of mobility and function.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen P Sayers, Ph.D., Principal Investigator — University of Missouri-Columbia School of Health Professions Physical Therapy Dept

IPD SHARING:
Plan to Share IPD: No